CLINICAL TRIAL: NCT05583448
Title: Post-market Clinical Follow-up Study of the ExploR™ Radial Head System (Implants and Instrumentation) - A Retrospective Enrollment/Prospective Follow-Up Consecutive Series Study
Brief Title: MDR ExploR Radial Head System PMCF
Status: Enrolling by invitation | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-77E
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Elbow Injury
MeSH Terms: conditions — Elbow Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- ExploR Radial Head: Subjects who have received the ExploR Radial Head Device.
  Interventions: Device: ExploR Radial Head

INTERVENTIONS:
Device: ExploR Radial Head — Patient must have undergone primary elbow arthroplasty with the ExploR Radial Head System according to a cleared indication.

SUMMARY:
The objective of this retrospective and prospective consecutive series PMCF study is to collect long-term data confirming safety, performance and clinical benefits of the ExploR Radial Head System (implants and instrumentation) when used for radial head arthroplasty.

DETAILED DESCRIPTION:
This is a global, multi-center, retrospective enrollment, prospective follow-up, consecutive series post-market clinical follow-up study. The intent of the study is that subjects who have already had the surgical implant will be retrospectively enrolled in the study and data will be collected for a minimum of 10 years post-operatively. Subjects treated with the device will be identified and invited to participate in the study. 93 subjects will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

Patient must have undergone primary elbow arthroplasty with the ExploR Radial Head System according to a cleared indication, which includes the following:

* Replacement of the radial head for degenerative or post-traumatic disabilities presenting pain, crepitation and decreased motion at the radio-humeral and/or proximal radio-ulnar joint with:

Joint destruction and/or subluxation visible on x-ray Resistance to conservative treatment

* Primary replacement after fracture of the radial head
* Symptomatic sequelae after radial head resection Patient must be 18 years of age or older. Patient must be willing and able to follow directions.

Exclusion Criteria:

* Infection
* Sepsis
* Osteomyelitis
* Uncooperative patient or patient with neurological disorders who are incapable of following directions
* Osteoporosis
* Metabolic disorders which may impair bone formation
* Osteomalacia
* Distant foci of infections which may spread to implant site
* Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Patient is a prisoner.
* Patient is a current alcohol or drug abuser.
* Patient has a psychiatric illness or cognitive deficit that will not allow for proper informed consent
* Patient is known to be pregnant or breastfeeding.
* Patient is unwilling to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population should be a consecutive series of subjects implanted with the ExploR Radial Head System. The aim is to include 93 radial head arthroplasty procedures in the study.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2022-08-16 (Actual); Primary Completion 2026-08-16 (Estimated); Study Completion 2035-07-19 (Estimated)

PRIMARY OUTCOMES:
Device Survivorship | 10 years
  Measured by recording and analyzing the incidence and frequency of revisions, complications and adverse events. Survivorship is calculated with Kaplan Meier.
Device Safety | 10 years
  Assessed by recording frequency of adverse events during the length of the study.

SECONDARY OUTCOMES:
QuickDASH | 1, 3, 5, 7, and 10 years
  QuickDASH measures musculoskeletal pain and function of the arm. Higher scores indicate higher severity of disability.

CONTACTS AND LOCATIONS:
Locations (2):
- Norton Healthcare, Louisville, Kentucky, United States
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No